CLINICAL TRIAL: NCT05173077
Title: Hybrid-sensor Breath Analysis for Colorectal Cancer Screening (HYCOR)
Brief Title: Hybrid-sensor Breath Analysis for Colorectal Cancer Screening
Acronym: HYCOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Latvia (Other)
Collaborators: Universitaet Innsbruck (Other); University of Ulm (Other)
Responsible Party: Principal Investigator, Marcis Leja, Director, Institute of Clinical and Preventive Medicine, University of Latvia
Other Study IDs: 1.1.1.1/20/A/035
Record Dates: First submitted 2021-10-24; First posted 2021-12-29 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Cancer; Polyp of Colon
Keywords: Volatile organic compounds; Colorectal cancer; Breath testing
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Exhaled air samples being stored in specific adsorbent tubes. Plasma/serum samples for group stratification. Faecal samples for occult blood testing and microbiota analysis. Tissue samples for specific VOCs analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Colorectal cancer patients: Patients with histologically confirmed colorectal cancer (adenocarcinoma)
  Interventions: Device: Breath sampling for VOC detection; Other: Blood sample collection; Diagnostic Test: Microbiota testing
- Control group patients without colorectal cancer: Patients without colorectal malignant disease according to data obtained in colonoscopy
  Interventions: Device: Breath sampling for VOC detection; Other: Blood sample collection; Diagnostic Test: Microbiota testing; Diagnostic Test: Colonoscopy
- Average risk population: Average risk population of both genders aged 40-64 at the time of inclusion lacking alarm symptoms for gastrointestinal cancer
  Interventions: Other: Secondary validation study in general CRC screening settings; Other: Blood sample collection; Diagnostic Test: Microbiota testing; Diagnostic Test: Colonoscopy
- Colorectal cancer patients undergoing surgery: Patients with histologically confirmed colorectal cancer (adenocarcinoma) planned for surgical management
  Interventions: Procedure: Identification of specific VOCs in CRC tissue surgery material; Other: Blood sample collection; Diagnostic Test: Microbiota testing
- Patients with polyps undergoing polypectomy: Patients with colon polyps that will perform polypectomy
  Interventions: Device: Breath sampling for VOC detection; Other: Blood sample collection; Diagnostic Test: Microbiota testing; Diagnostic Test: Colonoscopy

INTERVENTIONS:
Procedure: Identification of specific VOCs in CRC tissue surgery material — Paired tissue samples will be taken during surgery for CRC. Tissue material from the same patient will be obtained from the cancerous tissue as well as from normal resected material without malignant infiltration. Minimum of 100 mg of each tissue per sample will be obtained. To compare the emission of VOCs in the CRC tissue surgery material to the emissions from normal tissue by GC-MS in a reasonable number of cancer cases.
  Groups: Colorectal cancer patients undergoing surgery
Other: Secondary validation study in general CRC screening settings — Altogether at least 1000 individuals relatively healthy 40-64 years old population-based collected individuals will get recruited. Breath samples will be collected by asking the study subjects to breath into hybrid breath analyser.
  To exclude significant colorectal lesions, laboratory-based FIT testing will be offered to the population cohort group for faecal occult blood in faeces. Serum and plasma samples will also be obtained to have them available if additional testing will be required. Individuals with a FIT test value over the cut-off value (>10 microg/g faeces) will be invited to colonoscopy. The data analysis procedures and classification models will be tested in this general population and cross-checked against FIT and colonoscopy results.
  Groups: Average risk population
Device: Breath sampling for VOC detection — Breath sampling will be performed by using a hybrid sensor device and or GC-MS analysis (by collecting breath samples in adsorbent tubes). Strict requirements for subjects will be imposed prior to the breath sampling to standardise the breath sampling and to limit the influence of confounding factors.
  Groups: Colorectal cancer patients; Control group patients without colorectal cancer; Patients with polyps undergoing polypectomy
Other: Blood sample collection — Serum, plasma sampling for group description and stratification.
Diagnostic Test: Microbiota testing — Faecal samples for microbiota testing.
Diagnostic Test: Colonoscopy — Colonoscopy will be used only according to the clinical indications.
  Groups: Average risk population; Control group patients without colorectal cancer; Patients with polyps undergoing polypectomy

SUMMARY:
The aim of this project is to promote the breath volatile marker concept for colorectal cancer (CRC) screening by advancing developing the application of a novel hybrid analyzer for the purpose.

The hybrid analyzer concept is expected to benefit of combining metal-oxide (MOX) and infrared spectrum (IR) sensor acquired data. The current study will be the first globally to address this concept in CRC detection. In addition, traditional methods, in particular, gas chromatography coupled to mass spectrometry (GC-MS) will be used to address the biological relevance of the VOCs emission from cancer tissue and will assist in further advances of the hybrid-sensing approach.

DETAILED DESCRIPTION:
For addressing the aims of the project, four specific research objectives have been set:

1. To identify cancer-related VOCs emitted by the CRC tissue via the comparison of VOCs emitted from cancer tissue with VOCs emitted by non-cancerous tissue (ex vivo surgery material) by GC-MS.
2. To identify the VOCs differentiating human breath from CRC patients and controls (by GC-MS) as well as compare the chemical signature of CRC patients' breath to the chemical signature of cancer tissue.
3. To evaluate the performance of the set of sensors in the hybrid analyzer and the performance of particular sensors for detecting CRC; to develop and validate a mathematical model for CRC detection.
4. To validate the hybrid analyzer in real-life CRC screening settings, i.e. versus the generally accepted CRC screening approach of faecal occult blood detection.
5. To compare faecal microbiome between CRC group and control.

The scientific results to be obtained during the current project are expected to elucidate the origin and metabolism of volatile biomarkers of CRC. This achievement, in turn, will facilitate the implementation of a new screening test based on the newly developed hybrid analyser into medical practice.

Identification of the VOCs patterns by the sensor array for CRC patients when compared to controls. Addressing these objectives will allow an in-depth understanding of the physiological background for exhaled VOCs in CRC patients and facilitate the development of technologies able to identify the disease and its precursors from an exhaled breath sample.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals (>18 years of age)
* Having signed the consent form
* Willingness to collaborate
* Able to provide a breath sample

  * For the cancer group: colorectal adenocarcinoma has to be documented histologically (histological diagnosis following gastric surgery is also accepted) or patients being confirmed adenocarcinoma during the course of the study.
  * For the non-cancer group: control group - any patient who have medical indications for a colonoscopy

Exclusion Criteria:

* The patient has not signed the consent form
* Patients who have had a complete bowel cleansing
* Other active malignancies
* Neoadjuvant chemotherapy, radiation therapy is currently underway
* Acute conditions (emergency surgery for the patient)
* Small bowel resection in the past
* Terminal renal failure (Chronic renal failure stage 4)
* Type I diabetes
* Bronchial asthma (active)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patient group: patients with known or suspected colorectal adenocarcinoma being admitted to the major specialized cancer centre in Latvia for diagnostic purpose, medical or surgical management will get recruited.
  Control group patients will be recruited in the major specialized endoscopy centre (Digestive Diseases Centre "GASTRO") in Latvia.
  Average m risk population: average risk population of both genders aged 40-64 at the time of inclusion lacking alarsymptoms for gastrointestinal cancer will get recruited. Those will be invited actively from the GP registries or registry of the National Health Services (the regulatory approval for this approach is already available). An equal proportion between the genders will be targeted.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Characteristic VOC pattern identification for colorectal cancer detection | 2 years following initiation of patient recruitment
  The characteristic VOC pattern based on sensor analysis and its performance indicators will be detected.
Specific chemistry identification in the exhaled breath | 2 years following initiation of patient recruitment
  Identification of specific chemistries (GC-MS analysis) originating from colorectal cancer. Volatiles will be separated using an Rt-Q-BOND column working in a constant flow of helium. The column temperature program will be optimized toward detection of observed volatiles. The SCAN, will be used for the untargeted analysis and identification of compounds of breath samples as well as for the quantification of more abundant species. Peak integration will be based on extracted ion chromatograms. The identification of compounds will be performed in two steps. The peak spectrum will be checked against the NIST mass spectral library. The NIST identification will be confirmed by comparing the respective retention times with retention times obtained on the basis of standard mixtures prepared from pure compounds. Whenever possible the VOC emission will be quantified using calibration mixtures prepared from pure liquid or gaseous substances.

SECONDARY OUTCOMES:
Identification of the best-performing sensors | 3 years following initiation of patient recruitment
  Decision on the optimal set of breath sensors that potentially will be included in a sensor analyser for CRC detection. Comparative analysis between the performance of different sensor performance in target disease identification.
Gut microbiota analysis in relation to breath VOCs | 3 years following initiation of patient recruitment
  Analysis of the role of faecal microbiota in the origin of VOCs in the exhaled breath.

OTHER OUTCOMES:
Confounding factor analysis | 3 years following initiation of patient recruitment
  The role of confounding factors will be addressed to address their role in VOC emission.
  Strict requirements for subjects will be imposed prior to the breath sampling to limit the influence of confounding factors. These will include i.a.; overnight fast (min 12h), refraining from smoking at least 2 hours prior to the sampling, refraining from alcohol consumption (1 day before sampling), avoiding excessive physical activity 1 hour prior to testing and refraining of using breath mints/chewing gums on the day of test.
  End-tidal portion of exhalation will be collected using buffered, or CO2 controlled sampling. Breath samples will be pre-concentrated using the sorbent tubes and stored at -86℃. An effort will be made to limit the storage time to 2 month. Next, samples will be analysed using GC-MS.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Latvia, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Result] Jurs PC, Bakken GA, McClelland HE. Computational methods for the analysis of chemical sensor array data from volatile analytes. Chem Rev. 2000 Jul 12;100(7):2649-78. doi: 10.1021/cr9800964. No abstract available. PMID 11749299
- [Result] van Keulen KE, Jansen ME, Schrauwen RWM, Kolkman JJ, Siersema PD. Volatile organic compounds in breath can serve as a non-invasive diagnostic biomarker for the detection of advanced adenomas and colorectal cancer. Aliment Pharmacol Ther. 2020 Feb;51(3):334-346. doi: 10.1111/apt.15622. Epub 2019 Dec 20. PMID 31858615
- [Result] Zhou W, Tao J, Li J, Tao S. Volatile organic compounds analysis as a potential novel screening tool for colorectal cancer: A systematic review and meta-analysis. Medicine (Baltimore). 2020 Jul 2;99(27):e20937. doi: 10.1097/MD.0000000000020937. PMID 32629696
- [Result] Sonoda H, Kohnoe S, Yamazato T, Satoh Y, Morizono G, Shikata K, Morita M, Watanabe A, Morita M, Kakeji Y, Inoue F, Maehara Y. Colorectal cancer screening with odour material by canine scent detection. Gut. 2011 Jun;60(6):814-9. doi: 10.1136/gut.2010.218305. Epub 2011 Jan 31. PMID 21282130
- [Result] Konvalina G, Haick H. Effect of humidity on nanoparticle-based chemiresistors: a comparison between synthetic and real-world samples. ACS Appl Mater Interfaces. 2012 Jan;4(1):317-25. doi: 10.1021/am2013695. Epub 2011 Dec 15. PMID 22121824
- [Result] Hagemann LT, Ehrle S, Mizaikoff B. Optimizing the Analytical Performance of Substrate-Integrated Hollow Waveguides: Experiment and Simulation. Appl Spectrosc. 2019 Dec;73(12):1451-1460. doi: 10.1177/0003702819867342. Epub 2019 Aug 22. PMID 31397586
- [Result] Hagemann LT , McCartney MM , Fung AG , Peirano DJ , Davis CE , Mizaikoff B . Portable combination of Fourier transform infrared spectroscopy and differential mobility spectrometry for advanced vapor phase analysis. Analyst. 2018 Nov 19;143(23):5683-5691. doi: 10.1039/c8an01192c. PMID 30232480
- [Result] Tutuncu E, Nagele M, Becker S, Fischer M, Koeth J, Wolf C, Kostler S, Ribitsch V, Teuber A, Groger M, Kress S, Wepler M, Wachter U, Vogt J, Radermacher P, Mizaikoff B. Advanced Photonic Sensors Based on Interband Cascade Lasers for Real-Time Mouse Breath Analysis. ACS Sens. 2018 Sep 28;3(9):1743-1749. doi: 10.1021/acssensors.8b00477. Epub 2018 Aug 20. PMID 30074387
- [Result] Glockler J, Jaeschke C, Kocaoz Y, Kokoric V, Tutuncu E, Mitrovics J, Mizaikoff B. iHWG-MOX: A Hybrid Breath Analysis System via the Combination of Substrate-Integrated Hollow Waveguide Infrared Spectroscopy with Metal Oxide Gas Sensors. ACS Sens. 2020 Apr 24;5(4):1033-1039. doi: 10.1021/acssensors.9b02554. Epub 2020 Mar 31. PMID 32189494
- [Result] Chandrapalan S, Arasaradnam RP. Urine as a biological modality for colorectal cancer detection. Expert Rev Mol Diagn. 2020 May;20(5):489-496. doi: 10.1080/14737159.2020.1738928. Epub 2020 Mar 11. PMID 32130868
- [Result] Gasenko E, Leja M, Polaka I, Hegmane A, Murillo R, Bordin D, Link A, Kulju M, Mochalski P, Shani G, Malfertheiner P, Herrero R, Haick H. How do international gastric cancer prevention guidelines influence clinical practice globally? Eur J Cancer Prev. 2020 Sep;29(5):400-407. doi: 10.1097/CEJ.0000000000000580. PMID 32740165
- [Result] Lawler M, Alsina D, Adams RA, Anderson AS, Brown G, Fearnhead NS, Fenwick SW, Halloran SP, Hochhauser D, Hull MA, Koelzer VH, McNair AGK, Monahan KJ, Nathke I, Norton C, Novelli MR, Steele RJC, Thomas AL, Wilde LM, Wilson RH, Tomlinson I; Bowel Cancer UK Critical Research Gaps in Colorectal Cancer Initiative. Critical research gaps and recommendations to inform research prioritisation for more effective prevention and improved outcomes in colorectal cancer. Gut. 2018 Jan;67(1):179-193. doi: 10.1136/gutjnl-2017-315333. PMID 29233930
- [Result] Broza YY, Mochalski P, Ruzsanyi V, Amann A, Haick H. Hybrid volatolomics and disease detection. Angew Chem Int Ed Engl. 2015 Sep 14;54(38):11036-48. doi: 10.1002/anie.201500153. Epub 2015 Jul 31. PMID 26235374